CLINICAL TRIAL: NCT06341257
Title: Efficacy and Toxicity of Stereotactic Central/Core Ablative Radiation Therapy (SCART) - A Prospective Observational Study
Brief Title: Efficacy and Toxicity of SCART
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participant
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, Hao-Shen Cheng, Attending Physician, Taichung Veterans General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VGHTCCTC_SCART001
Record Dates: First submitted 2024-03-21; First posted 2024-04-02 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Tumor Size Greater Than or Equal to 5 cm
Keywords: Bulky tumor; Palliative radiotherapy; Stereotactic Central/Core Ablative Radiation Therapy; Efficacy; Toxicity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SCART (Experimental): The patient will receive a dose of 21 Gy in 3 fractions, with the dose maintained at 5 Gy per fraction for the entire tumor GTV boundary.
  Interventions: Radiation: Stereotactic Central/Core Ablative Radiation Therapy (SCART)

INTERVENTIONS:
Radiation: Stereotactic Central/Core Ablative Radiation Therapy (SCART) — The patient will receive a dose of 21 Gy in 3 fractions, with the dose maintained at 5 Gy per fraction for the entire tumor GTV boundary.

SUMMARY:
This study is expected to enroll patients for a period of five years, with a total of 30 participants. It is a prospective observational study involving cancer patients with tumors having a longest diameter greater than or equal to 5 cm. Systemic drug therapy may be administered concurrently. The following inclusion criteria must be met for participation in the study: age greater than or equal to 18 years, Eastern Cooperative Oncology Group (ECOG) score ≤ 2, pathological confirmation of cancer diagnosis, tumor with a maximum diameter greater than or equal to 5 cm, one or more lesions, not suitable for surgery, patient has provided informed consent, patient receives SCART, and reproductive-age women must agree to take adequate contraceptive measures during the study and for six months after discontinuation of medication. The patient will receive a dose of 21 Gy in 3 fractions, with the dose maintained at 5 Gy per fraction for the entire tumor gross target volume (GTV) boundary. For certain patients, an additional two fractions of 5 Gy each were added using Stereotactic Body Radiotherapy (SBRT), resulting in a total dose of 5 Gy × 5 for the GTV boundary.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* ECOG score ≤ 2, pathological confirmation of cancer diagnosis
* Pathologically proved malignant tumor with a maximum diameter greater than or equal to 5 cm
* One or more lesions, not suitable for surgery
* Patient has provided informed consent

Exclusion Criteria:

* Pregnant
* Life expectancy less than six months
* Uncontrolled angina, arrythmia, and congestive heart failure
* History of malignant pleural effusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2025-04-08 (Actual)

PRIMARY OUTCOMES:
Local Control (LC) | From date of radiotherapy until the date of first documented progression, assessed up to 60 months
  a tumor volume equal to or less than the tumor volume at start of radiotherapy
Progression-Free Survival (PFS) | From date of radiotherapy until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  the time from inclusion to disease progression or death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lo SS, Fakiris AJ, Chang EL, Mayr NA, Wang JZ, Papiez L, Teh BS, McGarry RC, Cardenes HR, Timmerman RD. Stereotactic body radiation therapy: a novel treatment modality. Nat Rev Clin Oncol. 2010 Jan;7(1):44-54. doi: 10.1038/nrclinonc.2009.188. Epub 2009 Dec 8. PMID 19997074